CLINICAL TRIAL: NCT03558997
Title: A Study To Evaluate The Efficacy Of Dupilumab As An Adjunct For Subcutaneous Grass Immunotherapy To Reduce Provoked Allergic Rhinitis Symptoms Using The Nasal Allergen Challenge Model
Brief Title: Dupilumab As An Adjunct For Subcutaneous Grass Immunotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R668-ALG-16115
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Results first posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Experimental): Participants received placebo matched to Dupilumab and placebo matched to Timothy grass subcutaneous immunotherapy (SCIT) every 2 weeks (Q2W) for 16 weeks. Both placebo doses were administered with a gap of 1 or 7 days.
  Interventions: Drug: Placebo matching dupilumab; Drug: Placebo matching SCIT
- Dupilumab (Experimental): Participants received placebo matched to SCIT and subcutaneous (SC) injections of Dupilumab at a loading dose of 600 milligrams (mg) on Day 1, followed by a 300 mg for Q2W for 16 weeks. Both placebo matched to SCIT and Dupilumab doses were administered with a gap of 1 or 7 days.
  Interventions: Drug: Dupilumab; Drug: Placebo matching SCIT
- SCIT (Experimental): Participants received SCIT titrated up to a 4000 bioequivalent allergy unit (BAU) for 8 weeks followed by maintenance dose of 4000 BAU for following 8 weeks and SC injections of placebo matched to Dupilumab Q2W for 16 weeks. Both SCIT and placebo matched to Dupilumab doses were administered with a gap of 1 or 7 days.
  Interventions: Drug: Timothy Grass SCIT; Drug: Placebo matching dupilumab
- Dupilumab + SCIT (Experimental): Participants received SC injections of Dupilumab at a loading dose of 600 mg on Day 1, followed by 300 mg Q2W for 16 weeks and SCIT titrated up to 4000 BAU for 8 weeks followed by maintenance dose of 4000 BAU for following 8 weeks. Both SCIT and Dupilumab doses were administered with a gap of 1 or 7 days.
  Interventions: Drug: Dupilumab; Drug: Timothy Grass SCIT

INTERVENTIONS:
Drug: Dupilumab — Dupilumab was administered SC in a single-use, pre-filled glass syringe
  Other Names: DUPIXENT®; REGN668; SAR231893
  Arms: Dupilumab; Dupilumab + SCIT
Drug: Timothy Grass SCIT — Timothy grass extract was administered SC.
  Arms: Dupilumab + SCIT; SCIT
Drug: Placebo matching dupilumab — Placebo matching dupilumab was prepared in the same formulation without the addition of protein
  Arms: Placebo; SCIT
Drug: Placebo matching SCIT — Placebo matching SCIT was prepared in the same formulation (SCIT diluent) without the addition of Timothy grass extract
  Arms: Dupilumab; Placebo

SUMMARY:
The primary objective is to assess whether 16 weeks of treatment with dupilumab as an adjunct to Timothy Grass Subcutaneous Immunotherapy (SCIT) improves upon the efficacy of Timothy Grass SCIT to reduce provoked allergic rhinitis symptoms, as measured by Total Nasal Symptom Score (TNSS) after nasal allergen challenge (NAC) with Timothy Grass extract at week 17.

The secondary objectives of the study are:

* To assess whether 16 weeks of treatment with dupilumab as compared to placebo reduces provoked allergic rhinitis symptoms, as measured by TNSS after nasal allergen challenge (NAC) with Timothy Grass extract
* To assess whether 16 weeks of treatment with dupilumab as compared to dupilumab + SCIT reduces provoked allergic rhinitis symptoms, as measured by TNSS after nasal allergen challenge (NAC) with Timothy Grass extract
* To assess changes in serum Timothy-grass-specific immunoglobulin G4 (IgG4), serum Timothy grass-specific immunoglobulin E (IgE), and ratio of serum Timothy Grass-specific IgG4 to IgE over 16 weeks of treatment with dupilumab + SCIT as compared to SCIT monotherapy
* To evaluate the safety and tolerability of 16 weeks of treatment with dupilumab as an adjunct to Timothy Grass SCIT

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female participants aged 18 to 55
2. History of grass pollen-induced seasonal allergic rhinitis
3. Grass pollen allergy confirmed by both:

   1. Positive skin prick test (SPT) with Timothy Grass extract (mean wheal diameter at least ≥5 mm greater than a negative control)
   2. Positive serum Timothy Grass-specific IgE (≥0.35KU/L)

Key Exclusion Criteria:

1. Significant rhinitis, sinusitis, outside of the grass pollen season
2. Any contraindications to SCIT (i.e, severe cardiovascular disease, malignancies, autoimmune disease, use of beta blocker, asthma severe enough to require chronic medication, acute infection)
3. Use of systemic corticosteroids within 4 weeks of screening visits or any NAC visits
4. Abnormal lung function as judged by the investigator
5. A clinical history of asthma requiring chronic medication such as regular inhaled corticosteroids for >4 weeks per year
6. History of significant recurrent sinusitis, defined as 3 episodes per year for the last 2 years, all of which required antibiotic treatment
7. History of chronic sinusitis (with or without nasal polyps)
8. Tobacco smoking (ANY) within the last year

Note: Other protocol defined inclusion/ exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (17):
- United States (12):
  - Regeneron Investigational Site, Los Angeles, California
  - Regeneron Investigational Site, Mountain View, California
  - Regeneron Investigational Site, Walnut Creek, California
  - Regeneron Investigational Site, Baltimore, Maryland
  - Regeneron Investigational Site, Andover, Massachusetts
  - Regeneron Investigational Site, North Dartmouth, Massachusetts
  - Regeneron Investigational Site, St Louis, Missouri
  - Regeneron Investigational Site, Bellevue, Nebraska
  - Regeneron Investigational Site, Portland, Oregon
  - Regeneron Investigational Site, East Providence, Rhode Island
  - Regeneron Investigational Site, Seattle, Washington
  - Regeneron Investigational Site, Madison, Wisconsin
- Canada (5):
  - Regeneron Investigational Site, Kingston, Ontario
  - Regeneron Investigational Site, Mississauga, Ontario
  - Regeneron Investigational Site, Ottawa, Ontario
  - Regeneron Investigational Site, Toronto, Ontario
  - Regeneron Investigational Site, Québec, Quebec

REFERENCES:
- [Derived] Wipperman MF, Gayvert KM, Atanasio A, Wang CQ, Corren J, Covarrubias A, Setliff I, Chio E, Laws E, Wolfe K, Harel S, Maloney J, Herman G, Orengo JM, Lim WK, Hamon SC, Hamilton JD, O'Brien MP. Differential modulation of allergic rhinitis nasal transcriptome by dupilumab and allergy immunotherapy. Allergy. 2024 Apr;79(4):894-907. doi: 10.1111/all.16001. Epub 2024 Jan 27. PMID 38279910
- [Derived] Kamal MA, Franchetti Y, Lai CH, Xu C, Wang CQ, Radin AR, O'Brien MP, Ruddy M, Davis JD. Pharmacokinetics and Concentration-Response of Dupilumab in Patients With Seasonal Allergic Rhinitis. J Clin Pharmacol. 2022 May;62(5):689-695. doi: 10.1002/jcph.2004. Epub 2022 Jan 6. PMID 34791679
- [Derived] Corren J, Saini SS, Gagnon R, Moss MH, Sussman G, Jacobs J, Laws E, Chung ES, Constant T, Sun Y, Maloney J, Hamilton JD, Ruddy M, Wang CQ, O'Brien MP. Short-Term Subcutaneous Allergy Immunotherapy and Dupilumab are Well Tolerated in Allergic Rhinitis: A Randomized Trial. J Asthma Allergy. 2021 Aug 16;14:1045-1063. doi: 10.2147/JAA.S318892. eCollection 2021. PMID 34429614

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 214 participants were screened for study eligibility at 17 study sites in United States and Canada, of whom 103 were randomized to receive the study treatment. Screen failure was mostly due to inclusion criteria not met/exclusion criteria met.
Pre-assignment Details: Participants who met the eligibility criteria were randomized in 1:1:1:1 ratio to 1 of 4 treatment groups: Placebo, Dupilumab, Subcutaneous immunotherapy (SCIT) and Dupilumab + SCIT.
Groups:
- Placebo: Participants received placebo matched to Dupilumab and placebo matched to Timothy grass subcutaneous immunotherapy (SCIT) every 2 weeks (Q2W) for 16 weeks. Both placebo doses were administered with a gap of 1 to 7 days.
- Dupilumab: Participants received placebo matched to SCIT and subcutaneous (SC) injections of Dupilumab at a loading dose of 600 milligrams (mg) on Day 1, followed by a 300 mg for Q2W for 16 weeks. Both placebo matched to SCIT and Dupilumab doses were administered with a gap of 1 to 7 days.
- SCIT: Participants received SCIT titrated up to a 4000 bioequivalent allergy unit (BAU) for 8 weeks followed by maintenance dose of 4000 BAU for following 8 weeks and SC injections of placebo matched to Dupilumab Q2W for 16 weeks. Both SCIT and placebo matched to Dupilumab doses were administered with a gap of 1 to 7 days.
- Dupilumab + SCIT: Participants received SC injections of Dupilumab at a loading dose of 600 mg on Day 1, followed by 300 mg Q2W for 16 weeks and SCIT titrated up to 4000 BAU for 8 weeks followed by maintenance dose of 4000 BAU for following 8 weeks. Both SCIT and Dupilumab doses were administered with a gap of 1 to 7 days.
Period: Overall Study
Arm/Group | Placebo | Dupilumab | SCIT | Dupilumab + SCIT
Started | 25 | 26 | 26 | 26
Completed | 24 | 24 | 18 | 24
Not Completed | 1 | 2 | 8 | 2
Not completed — Adverse Event | 0 | 2 | 5 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab | SCIT | Dupilumab + SCIT | Total
Number analyzed (Participants) | 25 | 26 | 26 | 26 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.6 (11.05) | 40.3 (11.19) | 37.8 (11.25) | 33.0 (10.58) | 36.5 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 14 | 10 | 50
  Male | 15 | 10 | 12 | 16 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5 | 1 | 11
  Not Hispanic or Latino | 21 | 24 | 21 | 25 | 91
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 3 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 4 | 2 | 12
  White | 20 | 18 | 17 | 21 | 76
  More than one race | 1 | 2 | 1 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2
Total nasal symptom score (TNSS) Area under Curve (AUC) [0-1 hour (hr)] at Baseline [Mean (Standard Deviation); unit: Score on a Scale*hour] — TNSS was a participant-reported composite symptom assessment of 4 symptoms (rhinorrhea, nasal congestion, nasal itching & sneezing) each scored on a scale from 0 to 3 where 0 = none, 3 = severe. TNSS total score was ranged from 0 to 12, where higher the score indicated more severe symptoms. AUC of TNSS/component from time of the first observation to time of the last observation (AUC [0-1 hour]) was calculated by using the trapezoid rule.
  Score on a Scale*hour | 5.34 (2.175) | 5.03 (2.193) | 4.66 (1.987) | 4.69 (1.720) | 4.93 (2.015)
Timothy Grass Pollen IgG4 [Median (Inter-Quartile Range); unit: Miligram per Liter (mg/L)] — Measurement of Timothy Grass specific IgG4 was performed in serum or plasma to determine effects on biomarkers of relevant physiological and pathogenic processes.
  Miligram per Liter (mg/L) | 0.080 [0.080 to 0.210] | 0.080 [0.080 to 0.170] | 0.080 [0.080 to 0.190] | 0.080 [0.080 to 0.210] | 0.080 [0.080 to 0.210]
Timothy Grass Specific Immunoglobulin E (sIgE) [Median (Inter-Quartile Range); unit: Kilo Unit per Liter (kU/L)] — Measurement of Timothy Grass specific sIgE was performed in serum or plasma to determine effects on biomarkers of relevant physiological and pathogenic processes.
  Kilo Unit per Liter (kU/L) | 9.640 [3.890 to 37.100] | 4.810 [1.800 to 17.600] | 10.300 [3.600 to 20.600] | 11.250 [3.010 to 17.700] | 9.180 [3.000 to 20.700]
Log Transformed Timothy Grass Pollen IgG4 vs sIgE ratio [Median (Inter-Quartile Range); unit: Ratio] — Biomarkers measured in serum or plasma to determine effects on biomarkers of relevant physiological and pathogenic processes.
  Ratio | -1.970 [-2.390 to -1.460] | -1.515 [-2.150 to -1.220] | -1.860 [-2.110 to -1.650] | -1.975 [-2.340 to -1.170] | -1.840 [-2.300 to -1.350]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Nasal Symptom Score (TNSS) Area Under Curve (AUC) (0-1 Hour (hr) Post Peak TNSS) in Response to Post Nasal Allergen Challenge (NAC) at Week 17
Description: TNSS was participant-reported composite symptom assessment of 4 symptoms (rhinorrhea, nasal congestion, nasal itching & sneezing), each scored on a scale from 0 to 3 where 0 = none, 3 = severe. TNSS total score was calculated as the sum of the response for all 4 individual nasal symptom scores and ranged from 0 to 12, where higher score indicated more severe symptoms. AUC of TNSS/component from time of the first observation to time of the last observation (AUC [0-1 hr]) was calculated by using the trapezoid rule. Data was reported for Dupilumab + SCIT and placebo matched to Dupilumab + SCIT monotherapy group in this outcome measure.
Time Frame: Baseline, Week 17
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | SCIT | Dupilumab + SCIT
Number analyzed (Participants) | 26 | 26
Percent Change | -56.76 (9.687) | -52.03 (8.462)
Statistical Analysis 1: Comparison: SCIT vs Dupilumab + SCIT; Test type: Superiority; p = 0.7185, ANCOVA; A Multiple imputation (MI) method addressed missing values in AUC (percent change from baseline) - Seeds: 16115 and 51161 with imputation size 40; Least Square (LS) Mean Difference = 4.73, 95% CI 2-sided [-21.023 to 30.487] — The confidence interval (CI) with p-value was based on treatment difference (Dupilumab + SCIT vs SCIT) of the LS mean using analysis of covariance (ANCOVA) model with baseline measurement as covariate and the treatment as fixed factor

2. Secondary Outcome: Change From Baseline in Total Nasal Symptom Score (TNSS) Area Under Curve (AUC) Post Nasal Allergen Challenge (NAC) Over the First Hour After the Challenge (0-1 Hour (hr) Post Peak TNSS) at Week 17 in SCIT vs. Dupilumab + SCIT
Description: TNSS was participant-reported composite symptom assessment of 4 symptoms (rhinorrhea, nasal congestion, nasal itching & sneezing) each scored on a scale from 0 to 3 where 0 = none, 3 = severe. TNSS total score was calculated as the sum of the response for all 4 individual nasal symptom scores and ranged from 0 to 12, where higher score indicated more severe symptoms. AUC of TNSS/component from time of the first observation to time of the last observation (AUC [0-1 hr]) was calculated by using the trapezoid rule. Data was reported for Dupilumab + SCIT and placebo matched to Dupilumab + SCIT monotherapy group in this outcome measure.
Time Frame: Baseline, Week 17
Population: FAS included all randomized participants. Efficacy analyses were based on the treatment allocated at randomization (as randomized).
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale*hour
Arm/Group | SCIT | Dupilumab + SCIT
Number analyzed (Participants) | 26 | 26
Score on a Scale*hour | -3.07 (0.361) | -2.77 (0.321)
Statistical Analysis 1: Comparison: SCIT vs Dupilumab + SCIT; Test type: Superiority; p = 0.5438, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square (LS) Mean Difference = 0.30, 95% CI 2-sided [-0.661 to 1.254] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Total Nasal Symptom Score (TNSS) Area Under Curve (AUC) Post Nasal Allergen Challenge (NAC) Over the First Hour After the Challenge (0-1 Hour (hr) Post Peak TNSS) at Week 17 in Placebo vs. Dupilumab
Description: TNSS was participant-reported composite symptom assessment of 4 symptoms (rhinorrhea, nasal congestion, nasal itching & sneezing) each scored on a scale from 0 to 3 where 0 = none, 3 = severe. TNSS total score was calculated as the sum of the response for all 4 individual nasal symptom scores and ranged from 0 to 12, where higher score indicated more severe symptoms. AUC of TNSS/component from time of the first observation to time of the last observation (AUC [0-1 hr]) was calculated by using the trapezoid rule. Data was reported for Dupilumab + placebo matched to SCIT and placebo matched to dupilumab + placebo matched to SCIT group in this outcome measure.
Time Frame: Baseline, Week 17
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale*hour
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 25 | 26
Score on a Scale*hour | -1.85 (0.323) | -1.83 (0.329)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; Test type: Superiority; p = 0.9559, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square (LS) Mean Difference = 0.03, 95% CI 2-sided [-0.877 to 0.928] — The confidence interval (CI) with p-value was based on treatment difference (Dupilumab vs Placebo) of the LS mean using analysis of covariance (ANCOVA) model with baseline measurement as covariate and the treatment as fixed factor

4. Secondary Outcome: Percent Change From Baseline in Total Nasal Symptom Score (TNSS) Area Under Curve (AUC) Post Nasal Allergen Challenge (NAC) Over the First Hour of the Challenge (0-1 Hour (hr) Post Peak TNSS) at Week 17
Description: TNSS was participant-reported composite symptom assessment of 4 symptoms (rhinorrhea, nasal congestion, nasal itching & sneezing) each scored on a scale from 0 to 3 where 0 = none, 3 = severe. TNSS total score was calculated as the sum of the response for all 4 individual nasal symptom scores and ranged from 0 to 12, where higher score indicated more severe symptoms. AUC of TNSS/component from time of the first observation to time of the last observation (AUC [0-1 hr]) was calculated by using the trapezoid rule. Data was reported for Dupilumab + placebo matched to SCIT and placebo matched to dupilumab + placebo matched to SCIT.
Time Frame: Baseline, Week 17
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 25 | 26
Percent Change | -28.82 (8.427) | -21.57 (8.415)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; Test type: Superiority; p = 0.5416, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square (LS) Mean Difference = 7.25, 95% CI 2-sided [-16.028 to 30.530] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Change From Baseline in TNSS Area Under Curve (AUC) Post Nasal Allergen Challenge (NAC) Over the First Hour of the Challenge (0-1 Hour (hr) Post Peak TNSS) at Week 17
Description: TNSS was participant-reported composite symptom assessment of 4 symptoms (rhinorrhea, nasal congestion, nasal itching & sneezing) each scored on a scale from 0 to 3 where 0 = none, 3 = severe. TNSS total score was calculated as the sum of responses for all 4 individual nasal symptom scores and ranged from 0 to 12, where higher score indicated more severe symptoms. AUC of TNSS/component from time of the first observation to time of the last observation (AUC [0-1 hr]) was calculated by using the trapezoid rule. Data was reported for Dupilumab + SCIT and Dupilumab + placebo matched to SCIT group in this outcome measure.
Time Frame: Baseline, Week 17
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale*hour
Arm/Group | Dupilumab | Dupilumab + SCIT
Number analyzed (Participants) | 26 | 26
Score on a Scale*hour | -1.83 (0.329) | -2.77 (0.321)
Statistical Analysis 1: Comparison: Dupilumab vs Dupilumab + SCIT; Test type: Superiority; p = 0.0414, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square (LS) Mean Difference = -0.94, 95% CI 2-sided [-1.848 to -0.037] — The confidence interval (CI) with p-value was based on treatment difference (Dupilumab + SCIT vs Dupilumab) of LS mean difference using analysis of covariance (ANCOVA) model with baseline measurement as covariate and the treatment as fixed factor

6. Secondary Outcome: Percent Change From Baseline in TNSS Area Under Curve (AUC) Post Nasal Allergen Challenge (NAC) Over the First Hour of the Challenge (0-1 Hour (hr) Post Peak TNSS) at Week 17
Description: TNSS was participant-reported composite symptom assessment of 4 symptoms (rhinorrhea, nasal congestion, nasal itching & sneezing) each scored on a scale from 0 to 3 where 0 = none, 3 = severe. TNSS total score was calculated as the sum of the response for all 4 individual nasal symptom scores and ranged from 0 to 12, where higher score indicated more severe symptoms. AUC of TNSS/component from time of the first observation to time of the last observation (AUC [0-1 hr]) was calculated by using the trapezoid rule. Data was reported for Dupilumab + SCIT and Dupilumab + placebo matched to SCIT group in this outcome measure.
Time Frame: Baseline, Week 17
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Dupilumab | Dupilumab + SCIT
Number analyzed (Participants) | 26 | 26
Percent Change | -21.57 (8.415) | -52.03 (8.462)
Statistical Analysis 1: Comparison: Dupilumab vs Dupilumab + SCIT; Test type: Superiority; p = 0.0108, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square (LS) Mean Difference = -30.45, 95% CI 2-sided [-53.874 to -7.034] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Change From Baseline in Serum Timothy Grass Specific Immunoglobulin G4 (sIgG4) to Week 17
Description: Measurement of Timothy Grass specific IgG4 was performed in serum or plasma to determine effects on biomarkers of relevant physiological and pathogenic processes. Data was reported for Dupilumab + SCIT and placebo matched to Dupilumab + SCIT monotherapy group in this outcome measure. Missing values were imputed by Last Observation Carried Forward (LOCF) method for visits between post-baseline to Week 17.
Time Frame: Baseline, Week 17
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Milligram per Liter (mg/L)
Arm/Group | SCIT | Dupilumab + SCIT
Number analyzed (Participants) | 26 | 26
Milligram per Liter (mg/L) | 1.705 [0.520 to 6.090] | 3.550 [0.630 to 8.250]
Statistical Analysis 1: Comparison: SCIT vs Dupilumab + SCIT; Test type: Superiority; p = 0.1449, ANCOVA; Median Difference = 0.665, 95% CI 2-sided [-0.770 to 3.2100] — P-value was based on treatment differences of median change using rank based ANCOVA model with baseline measurement as covariate & treatment as fixed factors. Median difference & its 95% CI estimated with Hodges-Lehmann method

8. Secondary Outcome: Percent Change From Baseline in Serum Timothy Grass Specific Immunoglobulin G4 (sIgG4) to Week 17
Description: Measurement of Timothy Grass specific IgG4 was performed in serum or plasma to determine effects on biomarkers of relevant physiological and pathogenic processes. Data was for Dupilumab + SCIT and placebo matched to Dupilumab + SCIT monotherapy group in this outcome measure. Missing value was imputed by LOCF method for visits between post-baseline to Week 17.
Time Frame: Baseline, Week 17
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | SCIT | Dupilumab + SCIT
Number analyzed (Participants) | 26 | 26
Percent Change | 1444.49 [650.00 to 2650.00] | 1896.25 [700.00 to 5050.00]
Statistical Analysis 1: Comparison: SCIT vs Dupilumab + SCIT; Test type: Superiority; p = 0.1231, ANCOVA; Median Difference = 335.3, 95% CI 2-sided [-551.47 to 1746.55] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Change From Baseline in Serum Timothy Grass Specific Immunoglobulin E (sIgE) to Week 17
Description: Measurement of Timothy Grass specific sIgE was performed in serum or plasma to determine effects on biomarkers of relevant physiological and pathogenic processes. Data was reported for Dupilumab + SCIT and placebo matched to Dupilumab + SCIT monotherapy group in this outcome measure. Missing value was imputed by LOCF method for visits between post-baseline to Week 17.
Time Frame: Baseline, Week 17
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Kilo Unit per Liter (kU/L)
Arm/Group | SCIT | Dupilumab + SCIT
Number analyzed (Participants) | 26 | 26
Kilo Unit per Liter (kU/L) | 6.460 [2.750 to 15.900] | -2.990 [-10.890 to -0.940]
Statistical Analysis 1: Comparison: SCIT vs Dupilumab + SCIT; Test type: Superiority; p < 0.0001, ANCOVA; Median Difference = -13.325, 95% CI 2-sided [-23.9400 to -8.3600] — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: Percent Change From Baseline in Serum Timothy Grass Specific Immunoglobulin E (sIgE) to Week 17
Description: as for outcome 9
Time Frame: Baseline, Week 17
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | SCIT | Dupilumab + SCIT
Number analyzed (Participants) | 26 | 26
Percent Change | 81.27 [21.27 to 179.41] | -56.44 [-68.00 to -37.20]
Statistical Analysis 1: Comparison: SCIT vs Dupilumab + SCIT; Test type: Superiority; p < 0.0001, ANCOVA; Median Difference = -134.6, 95% CI 2-sided [-205.51 to -94.98] — [estimate comment as in outcome 7, analysis 1]

11. Secondary Outcome: Change From Baseline in Log-Transformed Value of Serum Timothy Grass Specific Immunoglobulin G4 (sIgG4) to Serum Timothy Grass Specific Immunoglobulin E (sIgE) Ratio to Week 17
Description: Biomarkers measured in serum or plasma to determine effects on biomarkers of relevant physiological and pathogenic processes. Data was reported for Dupilumab + SCIT and placebo matched to Dupilumab + SCIT monotherapy group in this outcome measure. Missing value was imputed by LOCF method for visits between post-baseline to Week 17.
Time Frame: Baseline, Week 17
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | SCIT | Dupilumab + SCIT
Number analyzed (Participants) | 26 | 26
Ratio | 0.745 [0.210 to 1.400] | 1.720 [1.360 to 2.130]
Statistical Analysis 1: Comparison: SCIT vs Dupilumab + SCIT; Test type: Superiority; p < 0.0001, ANCOVA; Median Difference = 0.840, 95% CI 2-sided [0.4500 to 1.2700] — [estimate comment as in outcome 7, analysis 1]

12. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) that developed or worsened or became serious during on-treatment period (time from the first dose of study drug up to the end of study [Week 24]). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-participant hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Baseline through Week 24
Population: The safety analysis set (SAF) included all randomized participants who received at least one injection of study drug, it was based on the treatment received (as treated).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab | SCIT | Dupilumab + SCIT
Number analyzed (Participants) | 25 | 26 | 26 | 26
Participants
  Participants with TEAEs | 21 | 18 | 24 | 22
  Participants with Serious TEAEs | 1 | 1 | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from the time the informed consent was signed until the participant's last study visit, regardless of seriousness or relationship to investigational product.Treatment-emergent adverse events were reported for the 16-week treatment period and the 8-week follow-up period.
Description: Reported AEs are treatment-emergent adverse events, which are defined as those that are not present at baseline or represent the exacerbation of a pre-existing condition during the treatment emergent period. The safety analysis set (SAF) included all randomized participants who received any study drug; it was based on the treatment received (as treated). The safety analyses were based on the SAF.
Arm/Group | Placebo | Dupilumab | SCIT | Dupilumab + SCIT
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/26 | 1/26 | 2/26
Other Adverse Events (participants affected / at risk) | 19/25 | 16/26 | 23/26 | 20/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Dupilumab (N=26) | SCIT (N=26) | Dupilumab + SCIT (N=26)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Dupilumab (N=26) | SCIT (N=26) | Dupilumab + SCIT (N=26)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site bruising (General disorders) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
Injection site erythema (General disorders) | 1 (3) | 1 (1) | 2 (5) | 4 (8)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 5 (37) | 4 (35)
Injection site pruritus (General disorders) | 1 (2) | 0 (0) | 4 (12) | 3 (12)
Injection site reaction (General disorders) | 8 (56) | 8 (64) | 11 (119) | 16 (342)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 3 (14) | 2 (16)
Injection site urticaria (General disorders) | 1 (2) | 0 (0) | 3 (12) | 2 (4)
Local reaction (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 4 (5) | 8 (11)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (9) | 5 (5) | 1 (1) | 10 (11)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 4 (4) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 3 (10) | 1 (4) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT03558997/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT03558997/SAP_001.pdf